CLINICAL TRIAL: NCT03447886
Title: Understanding Barriers to Initiation and Adherence to Adjuvant Endocrine Therapy in Young Breast Cancer Survivors of Diverse Racial, Ethnic, and Socio-economic Backgrounds: The EMPOWER Study
Brief Title: Understanding Barriers to Initiation and Adherence to Endocrine Therapy in Young Breast Cancer Survivors of Diverse Backgrounds
Status: Completed | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Rachel Freedman, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 17-581; U54CA156732 (NIH)
Record Dates: First submitted 2018-02-21; First posted 2018-02-27 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Quality Of Life: This study uses qualitative research methods, specifically semi-structured interviews.
  * This will include moderator guide development,
  * Phone interviews with breast cancer survivors will be conducted
  * Qualitative data analysis of the phone interviews will be conducted
  Interventions: Other: Phone interview

INTERVENTIONS:
Other: Phone interview — Collecting clinical and socio-demographic information.

SUMMARY:
The overall goal of this study is to qualitatively explore how behavioral, cultural, psychosocial, and economic barriers and facilitators affect the decision to start and adhere to endocrine therapy (ET) among young breast cancer survivors of diverse racial, ethnic, and socio-economic backgrounds with hormone receptor positive (HR+) breast cancer

DETAILED DESCRIPTION:
A qualitative study that will use interviews to gain an in depth understanding of factors affecting the decision to start and adhere to endocrine therapy (ET) among young breast cancer survivors of diverse racial, ethnic, and socio-economic backgrounds with hormone receptor positive (HR+) breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Are Hispanic, Latina, Black, or identify as socio-economically disadvantaged (any racial/ethnic background) as measured by an item of financial distress answering that they are "having difficulty paying the bills no matter what they do" to a question about their current household financial situation.18, 19
* report a history of Stage 1-3 breast cancer
* reports HR+ breast cancer and confirm that they have had a discussion with their doctor about adjuvant ET; OR indicate that they are taking ET, even if they do not know their HR status, answer they are HR-, or do not recall having a discussion about ET)
* not in active treatment (e.g., chemotherapy, radiation), with the exception of Herceptin
* at least 3 months, but no more than 3 years out of completion of active treatment
* no evidence of recurrent/metastatic disease
* at least 18, but< 45 years of age at diagnosis of first invasive breast cancer
* English or Spanish speaking
* are willing to consent to the interview

Exclusion Criteria:

* HR- breast cancer and indicate they are not taking ET
* HR+ breast cancer but do not confirm discussion of ET or indicate they are taking ET
* Stage 0 (DCIS) breast cancer
* Recurrent or metastatic disease
* Less than 3 months or more than 3 years post-active treatment
* Less than 18 years old or ≥45 years old at diagnosis

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women of all races
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2018-08-27 (Actual)

PRIMARY OUTCOMES:
Decision-making around endocrine therapy in young women with HR+ breast cancer. | 3 months-3 years post active treatment
  Open ended questions

SECONDARY OUTCOMES:
Barriers and challenges to endocrine therapy adherence | 3 months-3 years post active treatment
  Open ended questions
Social support | 3 months-3 years post active treatment
  Open ended questions
Health behaviors | 3 months-3 years post active treatment
  Open ended questions
Endocrine therapy adherence intervention preferences | 3 months-3 years post active treatment
  Open ended questions
Health literacy | 3 months-3 years post active treatment
  Brief Health Literacy Screener (Chew items)
Menopausal symptoms | 3 months-3 years post active treatment
  BCPT Symptom Checklist

CONTACTS AND LOCATIONS:
Overall Officials: Rachel A Freedman, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No